CLINICAL TRIAL: NCT06887387
Title: Application of Wearable Devices for Remote QT Interval Monitoring and Symptom Investigation for Patients With Long QT Syndrome
Brief Title: Wearable Devices for Patient Monitoring in Long QT Syndrome
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 173178
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable device — This is an observational study that does not impact routine clinical care for participants

SUMMARY:
The main research question of this study is whether wearable devices have utility in monitoring patients with Long QT syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Long QT Syndrome
* Aged 18 years or over
* Phone with iOS version 15 or Android OS 9.0 or higher
* Able and willing to provide informed consent

Exclusion Criteria:

* Unwilling or unable to give consent
* Ventricular pacing at recruitment
* Bundle branch block or pre-excitation at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of long QT syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
1. Determine the accuracy of repeated QT interval measurements using Fitbit-derived ECGs in patients with Long QT syndrome compared with the current standard (12-lead ECG and ambulatory monitors) | From enrollment to 3 months
2. Establish intra-patient QT variability from weekly Fitbit-ECGs and frequency of measurements over 500ms. | From enrollment to 3 months

SECONDARY OUTCOMES:
1. Establish the utility of wearable devices for determining symptom aetiology in LQTS. | From enrollment to 3 months
2. Develop pipelines for the analysis of ECG data collected remotely including use of in-house QT automated algorithms for future machine learning applications. | From enrollment to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William J Young, MBBS, PhD, Principal Investigator — Queen Mary University of London and St Bartholomew's Hospital
Locations (1):
- Barts and London Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No